CLINICAL TRIAL: NCT05165108
Title: Non-invasive Vagus Nerve Stimulation in the Treatment of Crohn's Disease - A Pilot Study
Acronym: VNS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Indiana University (Other)
Collaborators: ElectroCore INC (Industry)
Responsible Party: Principal Investigator, Sashidhar V. Sagi, Principal Investigator, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10734
Record Dates: First submitted 2021-09-07; First posted 2021-12-21 (Actual); Results first posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-02

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Non-Invasive VNS (Experimental): Non-Invasive VNS will decrease inflammation in people with Crohn's disease leading to decrease in inflammatory markers and symptoms of disease.
  Interventions: Device: Vagal Nerve Stimulator

INTERVENTIONS:
Device: Vagal Nerve Stimulator — A handheld device which consists of a battery powered portable stimulator with a digital control user interface that controls signal amplitude and two steel contact electrodes will deliver the nVNS electrical stimulation to the cervical Vagus nerve. The device has been approved by the U.S. Food and Drug Administration (FDA) for non-invasive Vagus nerve stimulator therapy for adjunctive use for the prevention and treatment of migraine and cluster headaches in adult patients.
  Other Names: GammaCore nVNS

SUMMARY:
To assess the safety and efficacy of transcutaneous vagal stimulation in adult patients with active Crohn's disease.

DETAILED DESCRIPTION:
Crohn's disease (CD) is a type of inflammatory bowel disease (IBD) characterized by chronic inflammation in the digestive tract. The pathogenesis of IBD involves immunological, genetic and environmental factors. Currently there is no cure for Crohn's disease and available medical and surgical treatments are expensive and often associated with significant side effects. Anti-tumor necrosis factor alpha (anti-TNF-α) agents are widely used for treatment of Crohn's disease. Electrical neuromodulation is a new treatment approach of bioelectronic medicine, involving molecular medicine, neuroscience, and bioengineering. Multiple possible mechanisms have been proposed for electrical neuromodulation in GI diseases, including central, autonomic, and/or enteric mechanisms. Vagal tone is significantly blunted in IBD and is associated with high TNF- α levels. Animal and preliminary human studies have demonstrated that electrical vagal nerve stimulation (VNS), including non-invasive vagal stimulation (nVNS), exerts an anti-inflammatory effect by harnessing the cholinergic anti-inflammatory pathway. In healthy humans nVNS has been shown to decrease tumor necrosis factor-α levels. Invasive VNS has been shown to improve inflammation in preliminary studies in patients with Crohn's disease.

Adult patients with active Crohn's disease will be asked to self-administer transcutaneous vagal nerve stimulation three times per day for 16 weeks. Inflammatory laboratory markers will be compared for each patient against their baseline levels to determine if the intervention helps reduce inflammation cause by their Crohn's disease. Questionnaires will be administered to evaluation their symptoms, and quality of life over the 16 week treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Crohn's disease diagnosis for at least 3 months, confirmed by clinical, biochemical, and endoscopic evaluations.
2. Patients with CD involving the small bowel and / or colon with active symptoms with Crohn's Disease Activity Index (CDAI) > 220 despite at least one conventional therapy (corticosteroids and/or immunosuppressives) with a stable dose will be included.
3. Elevated Fecal calprotectin ≥ 200 micro g/g within the past 4 weeks prior to enrollment
4. If on corticosteroids, the dose must be stable and ≤ 20mg/day prednisone or equivalent for at least 14 days before entry into study.
5. If on background immunosuppressive treatment the dose must be stable with the following parameters:
6. 56 days (8 weeks) for Immunomodulators (methotrexate, 6-MP, Azathioprine) and small molecules (upadacitinib)
7. 112 84 days (16 12 weeks) for biologics (Infliximab, Adalimumab, Vedolizumab, Ustekinumab, another biologic Risankizumab)
8. Clinical laboratory evaluations (including a chemistry panel, complete blood count [CBC], and urinalysis [UA]) within the reference range for the test laboratory, unless a typical consequence of CD or deemed not clinically significant by the Investigator.
9. Colonoscopy within the previous 1 year with no evidence of colonic dysplasia or cancer.
10. Able and willing to give written informed consent and comply with the requirements of the study protocol.

Exclusion Criteria:

1. Expectation to increase corticosteroids and/or immunosuppressive treatment
2. Presence of bowel stricture with pre-stenotic dilatation
3. Presence of intra-abdominal or perirectal abscess
4. Crohn's Disease Activity Index (CDAI) < 220
5. Fistula with clinical or radiological evidence of abscess
6. Perianal CD with or without rectal involvement
7. Ileostomy, colostomy, enteral or parenteral feeding
8. Short gut syndrome.
9. Clinical condition medically or surgically unstable that, at the discretion of the investigator would not be compatible with the patient's participation in the study
10. Any malignant neoplasia, in the year prior to screening ,except for nonmelanoma skin cancer.
11. Active treatment with antibiotics
12. Presence of active intestinal infection or documented infection by stool PCR or culture analysis in the previous 6 weeks
13. Continuous treatment with an anti-cholinergic medication, including over the counter medications.
14. Implantable electronic devices such as pacemakers, defibrillators, hearing aids, cochlear implants or deep brain stimulators.
15. Current tobacco or nicotine user within the past 4 weeks (to limit potential confounding effects of exposure to nicotine)
16. Bowel resection surgery within past 90 days prior to study enrollment and on no conventional IBD therapy, or planned surgery within the course of the study

18. Participation in any other Investigational drug and/or treatment currently or planned during the length of the study 19. Any condition which, in the opinion of the investigator, would jeopardize the subject's safety following exposure to a study intervention 20. Pregnancy or Lactation 21. Comorbid disease with high likelihood of requiring corticosteroid use 22. Inability to comply with study and follow-up procedures 23. Non-English speaking. 24. Known cardiac condition causing or with potential to cause arrhythmia 25. Patients diagnosed with narrowing of the arteries (carotid atherosclerosis) 26. Patients who have had surgery to cut the Vagus nerve in the neck (cervical vagotomy) 27. Patients with clinically significant untreated hypertension, hypotension, bradycardia, or tachycardia.

28. Have a metallic device such as a stent, bone plate or bone screw implanted at or near their neck.

29. Are using another device at the same time (e.g., TENS Unit, muscle stimulator)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2022-08-12 (Actual); Study Completion 2022-08-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sashidhar V Sagi, MD, Principal Investigator — Indiana University School of Medicine; Thomas V Nowak, MD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana University, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No
all IPD that underlie results in a publication

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Non-Invasive VNS
Started | 4
Completed | 2
Not Completed | 2

BASELINE CHARACTERISTICS:
Population: Adult patients with Crohn's disease
Arm/Group | Non-Invasive VNS
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.5 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in Fecal Calprotectin From Baseline to 16 Weeks
Description: This test can identify the level of inflammation in the colon of a person with Crohn's Disease. If a person diagnosed with Crohn's Disease subsequently shows low levels (50 -200 ug/mg) of fecal calprotectin, this means that the inflammation is being controlled, so the treatment regime is working.
Time Frame: Baseline and 16 weeks
Population: Data was only able to be collected from 1 participant at Week 16.
Measure: Mean (Standard Deviation); unit: ug/mg
Arm/Group | Non-Invasive VNS
Number analyzed (Participants) | 1
ug/mg | -102 (0)

2. Secondary Outcome: Change in Crohn's Disease Activity Index (CDAI) From Baseline to 16 Weeks
Description: CDAI range is minimum 0 and maximum 450. Zero is best score. Four hundred and fifty is the worst score. Lowering the CDAI score by 70 points or more is the goal for this study. A CDAI score of < or = 150 is considered remission.
Time Frame: Baseline and 16 Weeks
Population: Enrolled/Randomized patients
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Non-Invasive VNS
Number analyzed (Participants) | 2
score on a scale | 275.7 (.1)

3. Secondary Outcome: Change in Serum Cytokine Levels From Baseline to 16 Weeks
Description: Cytokine levels within the blood will be assessed and compared to baseline levels. The cytokines being assayed include C- reactive protein, tumor necrosis factor-alpha, Interferon-gamma, Transforming Growth Factor-beta and Interleukins (IL) - 1, 6, 10, 12, 17, 21, 23. (all cytokines will be presented at pg/mL)
Time Frame: 16 Weeks
Population: No data was collected for this endpoint. This outcome was not measured due to lack of funding available for the project.
Arm/Group | Non-Invasive VNS
Number analyzed (Participants) | 0

4. Secondary Outcome: Evaluating Change in HRV From Baseline Until Study Completion.
Description: Heart Rate Variability (HRV)
Time Frame: 16 Weeks
Population: No data was collected for this endpoint. Heart Rate Variability data was not made available to MD and staff because of staffing changes.
Arm/Group | Non-Invasive VNS
Number analyzed (Participants) | 0

5. Secondary Outcome: Change in Insulin Levels After First Stimulation
Description: Serum Insulin levels in the blood will be assessed and compared prior to stimulation, and at 20 minutes and 40 minutes after the stimulation. (presented as mCU/mL)
Time Frame: Baseline Visit
Population: No data was collected for this endpoint. This was not measured due to lack of funding for the project.
Arm/Group | Non-Invasive VNS
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Through study completion, approximately 16 weeks
Description: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Arm/Group | Non-Invasive VNS
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2024-02-01): https://cdn.clinicaltrials.gov/large-docs/08/NCT05165108/Prot_000.pdf